CLINICAL TRIAL: NCT03964259
Title: Pilot Study on the Reduced Intravenous Fluids to Improve Clearance of High-Dose Methotrexate (HDMTX) in Children With Lymphoma or Acute Lymphoblastic Leukemia
Brief Title: Reduced IV Fluids to Improve Clearance of HDMTX in Children w/Lymphoma or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-18-14244; NCI-2019-03468 (Other: NCI/CTRP)
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Lymphoma; Acute Lymphoblastic Leukemia; Pediatric Cancer; Pediatric ALL; Pediatric Lymphoma
Keywords: High Dose Methotrexate; HDMTX; Intravenous Fluids
MeSH Terms: conditions — Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: The study uses a prospective randomized controlled crossover study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Hydration Regimen (Active Comparator): In the standard intravenous fluid (IVF) protocol, following completion of HDMTX infusion, post HDMTX IVF will be initiated at 125 mL/m2/hr (no maximum mL/hr total rate).
  Interventions: Drug: Intravenous fluids
- Reduced hydration regimen (Experimental): The reduced intravenous fluid (IVF) protocol, post HDMTX IVF will be initiated at 62.5 mL/m2/hr following completion of HDMTX infusion.
  Interventions: Drug: Intravenous fluids

INTERVENTIONS:
Drug: Intravenous fluids — Administration of post HDMTX intravenous fluids (IVF)

SUMMARY:
To determine whether a reduced volume hydration regimen will lead to a shorter time to methotrexate clearance when compared to a standard intravenous (IV) hydration regimen.

DETAILED DESCRIPTION:
This study uses a prospective randomized controlled crossover study design. Neither patients nor clinicians are blinded to the standard versus reduced intravenous fluids (IVF) regimen. Patients are randomized to begin with standard volume or reduced volume IVF. Over the course of 4 cycles of High Dose Methotrexate (HDMTX), patients alternate between standard and reduced volume post hydration fluids protocols.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphoma or acute lymphoblastic leukemia
* Candidate for a minimum of 2 cycles HDMTX (5 g/m2) in the inpatient setting
* Creatinine clearance ≥ 65 mL/min by modified Schwartz equation
* Patients of childbearing potential must have a negative pregnancy test (serum or urine)
* Lactating female patients must agree not to nurse a child while on this trial
* All patients and/or their parents or legal guardians must provide written informed consent, with assent provided if applicable

Exclusion Criteria:

* Trisomy 21
* History of dialysis within 30 days prior to study registration or currently on dialysis
* Polyuric renal dysfunction
* Pregnancy
* Known or suspected pleural effusion
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Time elapsed (in hours) from end of HDMTX to a serum methotrexate level <0.1 micromol/L | 63 Days
  To determine whether a reduced volume hydration regimen will lead to a shorter time to methotrexate clearance when compared to a standard IV hydration regimen by measuring serum methotrexate levels twenty-four hours following the end of the high dose methotrexate ( HDMTX) infusion, and continuing every twelve hours until the methotrexate level is less than 0.1 micromol/L.

SECONDARY OUTCOMES:
Markers of kidney toxicity | 84 Days
  To determine the effect of a reduced volume hydration regimen on markers of kidney toxicity (nephrotoxicity) by evaluating serum creatinine levels from baseline levels as well as the maximum decrease in estimated glomerular filtration rate (GFR) utilizing the modified Schwartz equation, following each HDMTX cycle.
Markers of fluid overload | 84 Days
  To determine the effect of a reduced volume hydration regimen on markers of fluid overload by evaluating maximum weight gain during each hospitalization, and by evaluating the incidence of NCI Common Terminology Criteria for Adverse Events (CTCAE) version v5.0 ≥ grade 1 clinical sequelae of hydration such as facial edema, pulmonary edema, abdominal distension, extremity edema, and weight gain.
Effects on therapy delays | 84 Days
  To examine the effects of a reduced volume hydration regimen on treatment schedule by measuring the number of days subsequent therapy is delayed for reasons other than scheduling issues or preferences.
Effects on development of severe mucositis | 84 Days
  To examine the effects of a reduced volume hydration regimen on development of severe mucositis by measuring the incidence of grade ≥ 3 (CTCAE v5.0) mucositis.

CONTACTS AND LOCATIONS:
Overall Officials: Cady P Noda, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/ Massey Cancer Center/ Children's Hospital of Richmond, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noda C, Gwaltney L, Sabo R, Lo M, Schefft M. Standard Versus Reduced Hydration to Improve Elimination of High-Dose Methotrexate in Pediatric Patients: A Controlled Crossover Trial. Pediatr Blood Cancer. 2025 Apr;72(4):e31566. doi: 10.1002/pbc.31566. Epub 2025 Jan 27. PMID 39868759

DOCUMENTS (1):
  • Informed Consent Form (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT03964259/ICF_000.pdf